CLINICAL TRIAL: NCT04822103
Title: A Real-World Study Evaluating the Effectiveness and Safety of Immune Checkpoint Inhibitors and Chemotherapy for Advanced Esophageal Cancer
Brief Title: A Real-World Study of Immune Checkpoint Inhibitors and Chemotherapy for Advanced Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: The People's Hospital of Gaozhou (Other); The General Hospital of Southern Theater Command (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); First Affiliated Hospital of Shantou University Medical College (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Shantou Central Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RICE-retro
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; real-world study; immunotherapy; chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of preoperative chemotherapy as standard therapy is well-established for advanced esophageal cancer. Immunotherapeutic agents such as Immune checkpoint inhibitors has been shown to improve objective response rate in solid tumors. However, there is a paucity of data regarding the efficacy and safety of preoperative immunotherapy plus chemotherapy in esophageal cancer patients in real-world practice. This study set out to investigate whether the combination of preoperative chemotherapy and immune checkpoint inhibitors is beneficial to improve the objective response rate as well as the pathological complete response rate in a real-world scenario.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as esophageal squamous cell carcinoma
* KPS≥80
* Adequate organ function
* No distant metastasis
* The diseases could be resected or potentially resectable after immunochemotherapy assessed by a thoracic oncologist

Exclusion Criteria:

* incomplete medical record which affects statistical analysis
* have participated in previous interventional clinical trials
* other situations evaluated by investigators not meet the enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as potentially resectable (including initially-unresectable) esophageal squamous cell carcinoma via pathological specimen, KPS ≥ 80, has adequate organ function and no distant metastasis are included in the study
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 weeks
  Objective Response Rate
Safety as measured by number of participants with Grade 3 and 4 adverse events | Up to 12 weeks
  Number of Grade 3 and 4 adverse events as defined by CTCAE v5.0
Feasibility of immunochemotherapy defined as at least 80% of the patients completed all planned courses | Up to 36 weeks
  The feasibility of immunochemotherapy was defined as at least 80% of the patients completed all planned courses.

SECONDARY OUTCOMES:
Pathologic complete response rate (pCR) | Three to five working days after surgery
  The rate of pathologic complete response rate after the combined treatment of chemotherapy and immunotherapy following surgery
R0 resection rate | Three to five working days after surgery
  The R0 resection rate of esophagectomy
Overall survival | from the date of diagnosis to the date of death, assessed up to 100 months
  Overall survival rate
Event-free survival | from the date of treatment initiation to the date of first progression (local recurrence of tumor or distant metastasis) or death from any cause, assessed up to 100 months
  EFS
Major pathological response | Three to five working days after surgery
  ≤10% residual viable tumor follow NAIC

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong

REFERENCES:
- [Derived] Yang W, Ma SC, Fang Z, Liu Y, Zhang X, Wang F, Wang C, Wang Y, Wang X, Chen W, Luo H, Yang L, Zhang S, Zeng B, Liu Z, Ou Q, Cai J, Yeung SJ, Cheng C. TP53-centric ctDNA complements PET/CT for non-invasive assessment of pathological complete response and survival after neoadjuvant immunochemotherapy in esophageal squamous cell carcinoma: a prospective cohort study. Int J Surg. 2025 May 1;111(5):3256-3268. doi: 10.1097/JS9.0000000000002341. PMID 40146232